CLINICAL TRIAL: NCT02594943
Title: Endodrill vs. Conventional Biopsy. Evaluation of Diagnostic Capacity in Diffuse Gastric Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too narrow inclusion criteria. Impossible to recruit patients.
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Martin Jeremiasen, Consultant Surgeon, Region Skane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Endodrill II
Record Dates: First submitted 2015-10-27; First posted 2015-11-03 (Estimated); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Stomach Neoplasms
Keywords: Diagnostics; Biopsy; Diffuse gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Signet Ring Cell | interventions — Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Biopsy (Active Comparator): 4 out of 8 biopsies taken with a Boston Scientific Large capacity with needle biopsy forceps from the suspected tumor tissue in the stomach. They will be taken in random order "blinded" for the person performing the examination.
  Interventions: Device: Boston Scientific Large Capacity with needle Biopsy
- Endodrill Biopsy (Active Comparator): 4 out of 8 biopsies taken with the Endodrill 1A instrument from the suspected tumor tissue in the stomach. They will be taken in random order "blinded" for the person performing the examination.
  Interventions: Device: Endodrill 1A (BIBBInstruments, Lund, Sweden)

INTERVENTIONS:
Device: Boston Scientific Large Capacity with needle Biopsy — The investigators will use a conventional biopsy forceps for taking tissue biopsies in the GI tract. In a randomized order 4 out of total 8 biopsies will be taken with the conventional biopsy forceps from the tumor tissue.
  Arms: Conventional Biopsy
Device: Endodrill 1A (BIBBInstruments, Lund, Sweden) — The investigators will use the Endodrill, a new device for endoscopic tissue sampling in the GI tract. In a randomized order 4 out of total 8 biopsies will be taken with the Endodrill instrument from the tumor tissue.
  Arms: Endodrill Biopsy

SUMMARY:
Endodrill is a new instrument for biopsy sampling in the GI-channel. The purpose of this study is as follows:

* Compare the Endodrill instrument with conventional biopsy forceps in terms of ability to establish the correct diagnosis of diffuse gastric cancer based on collected biopsies from tumor tissue.

DETAILED DESCRIPTION:
Endodrill is a newly constructed biopsy tool for flexible endoscopic use. It uses a drilling motion within a casing to harvest solid biopsies from tissue through the biopsy channel of a conventional flexible endoscope. It was originally designed for sampling of tissue from submucosal lesions. The investigators´ first study of the instrument is now finished. Endodrill is safe to use and generates more submucosal tissue compared to biopsies with a conventional biopsy forceps.

In this study, the investigators want to compare the Endodrill instrument´s ability to obtain representative tissue samples from a group of patients diagnosed with or suspected diffuse gastric cancer. 20 patients will be enrolled for this study. For each patient the investigators will collect 8 biopsies, 4 biopsies each with conventional biopsy and the Endodrill instrument respectively. The order will be randomized for each patient. For each specific biopsy the investigator will choose a particular site on the suspected tumor tissue without knowing which instrument that will be used for the biopsy. This procedure will be repeated for all 8 biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or with an established diagnosis of diffuse gastric cancer who are capable of stating a formal consent to participate in the study.

Exclusion Criteria:

* Mental illness
* Extreme co-morbidity (ASA>3)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Highest proportion (number) of representative biopsies from tumors of diffuse gastric cancer | 24 months

SECONDARY OUTCOMES:
Amount of (mm2 and %) submucosal tissue within the biopsies. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan Johansson, SrConsultant, Principal Investigator — Region Skåne

IPD SHARING:
Plan to Share IPD: No